CLINICAL TRIAL: NCT03745014
Title: Randomized Trial Assessing the Clinical Impact of Fast Bacteria Identification and Phenotypic Antimicrobial Susceptibility Testing on Patients With Bacteremic Due to Gram-Negative Rods
Brief Title: Clinical Impact of Fast Phenotypic Antimicrobial Susceptibility Testing on Patients With Gram-Negative Rod Bacteremia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No sites identified with IRB approval
Sponsor: Accelerate Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ECP000002
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Gram-negative Bacteremia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pheno (Active Comparator)
  Interventions: Diagnostic Test: Accelerate Pheno
- Standard of Care (Active Comparator)
  Interventions: Diagnostic Test: Standard of Care

INTERVENTIONS:
Diagnostic Test: Accelerate Pheno — The Accelerate Pheno™ system and PhenoTest™ BC Kit is a fully-integrated in vitro diagnostic system. It is FDA-cleared to perform ID of bacteria and yeast in less than 90 minutes and AST in less than 7 hours, on average, directly from positive blood culture.
  Arms: Pheno
Diagnostic Test: Standard of Care — Standard blood culture work up as determined by the site's microbiology lab.
  Arms: Standard of Care

SUMMARY:
The FDA-cleared Accelerate Pheno™ System and PhenoTest™ Blood Culture (BC) Kit will be used to assess the workflow impact of fast identification (ID)/ antimicrobial susceptibility testing (AST) in the microbiology lab and in the quality of care in patients with Gram-negative rod (GNR) bacteremia. Blood culture work up will be randomized to one of two arms: the positive blood culture will either undergo fast ID and AST using the Accelerate Pheno™ System and PhenoTest™ BC Kit or processing per the site's standard of care (SOC) procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age) hospitalized patients with positive blood culture due to gram-negative rod (on Gram stain)
* Blood culture drawn in the Emergency Department (ED)

Exclusion Criteria:

* Patients not admitted to hospital
* Patients discharged from hospital prior to blood culture positivity
* Only the first positive blood culture for each patient of each hospitalization will be included during the study period; any subsequent episode of bloodstream infection (BSI) will be excluded
* Positive blood culture with GNR in the prior 7 days (if known at the time of randomization)
* Transferred from an outside hospital and had a history of a previously positive blood culture of the same organism in the prior 7 days (if known at the time of randomization)
* GNR plus gram-positive organism, gram-negative cocci, and/or yeast detected on blood culture Gram stain
* Deceased or palliative care at the time of randomization
* Patient who is moribund (does not survive the initial 72 hours after enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking (DOOR) - composite outcome | 30 days
  The primary endpoint is the probability that a patient will have a better DOOR when the Accelerate PhenoTest™ BC kit is used on positive blood cultures due to gram-negative rods compared to the standard of care